CLINICAL TRIAL: NCT04522934
Title: A Pilot Randomized, Controlled Trial of the Effectiveness of Pain Neuroscience Education on Pain Intensity, Patients' Attitudes and Beliefs About Pain, Disability and Quality of Life After Arthroscopic Rotator Cuff Repair
Brief Title: A Pilot Randomized Trial of Pain Neuroscience Education in the Rehabilitation After Arthroscopic Rotator Cuff Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica del Maule (Other)
Responsible Party: Principal Investigator, Jorge Fuentes, Principal investigator, Universidad Católica del Maule
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Neuroscience Rotator Cuff
Record Dates: First submitted 2020-08-16; First posted 2020-08-21 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Rotator Cuff Injuries
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to groups by using an online random generator. This procedure was conducted by an external assessor. The allocation concealment strategy included the use of sealed-opaque and consecutively numbered envelopes.
Who Masked: Outcomes Assessor
Masking Description: The assessor responsible for the outcome measures was blinded to the subjetc´s treatment assignment. The assessor was not present in the room while the treatment was delivered. He returned once the treatment was completed to perform the measurements.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Neuroscience Education (Experimental): Patients received 24 sessions, in a 8-week period, of multimodal physiotherapy along with four sessions of pain neuroscience education.
  Interventions: Behavioral: Pain Neuroscience Education
- Biomedical Education (Active Comparator): Patients received 24 sessions, in an 8-week period, of multimodal physiotherapy along with four sessions of biomedical education.
  Interventions: Behavioral: Biomedical Education

INTERVENTIONS:
Behavioral: Pain Neuroscience Education — Patients received 24 sessions, in an 8-week period, of multimodal physiotherapy (therapeutic heat, manual therapy and exercises) along with four sessions of pain neuroscience education. The latter was focused on the influence of psychosocial factors in the experience of pain, differences between acute and chronic pain and central-peripheral awareness.
  Arms: Pain Neuroscience Education
Behavioral: Biomedical Education — Patients received 24 sessions, in an 8-week period, of multimodal physiotherapy (therapeutic heat, manual therapy and exercises) along with four sessions of biomedical education. The latter was focused on the anatomy and pathomechanics of the shoulder.
  Arms: Biomedical Education

SUMMARY:
The aim of this study was to evaluate the effects of a 8-week pain neuroscience education programme compared to a biomedical education programme on the rehabilitation of patients who undergo arthroscopic rotator cuff repair. Outcome measures included pain intensity, patients' attitudes and beliefs about pain, disability and quality of life.

DETAILED DESCRIPTION:
This was a single-blinded, randomized parallel study. Twenty- nine patients who undergo arthroscopic rotator cuff repair took part in a multimodal physiotherapy programme and were allocated to two groups. Patients in the experimental group - PNE (n= 16) received multimodal physiotherapy along with pain neuroscience education, and the control group- PME (n=13) received multimodal physiotherapy along with biomedical education. The multimodal treatment included 1-hour sessions 3 times per week for 8 weeks (24 sessions). In addition, the education component (PNE, PME) consisted of 4 education sessions of 30 minutes duration, on a one-to-one basis, once per week at the start of the programme.

Physiotherapists involved in the delivery of the interventions were previously trained on both, the theoretical and practical aspects related to the protocols of multimodal physiotherapy and specially on the education component.

Outcome measures included pain intensity (pain intensity numerical rating score), catastrophizing, kinesiophobia, disability and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* People aged 30 to 59 years with shoulder pain for more than three months, with torn rotator cuff repaired by arthroscopy.

Exclusion Criteria:

* Subjects unable to understand, read or speak Spanish, or participated in a programme for psychological management of chronic pain, or presented with generalised pain.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-01-25 (Actual)

PRIMARY OUTCOMES:
Change Pain intensity: visual analogue scale | From baseline to the end of intervention (8 weeks)
  The visual analogue scales is a self-reporting measure of pain intensity. This involves asking patients to rate their pain intensity by selecting a point in a straight horizontal line of fixed length, usually 10 cm. The ends are defined as the extreme limits of the parameter to be measured orientated from the left (worst) to the right (best). The Minimal Clinically Important Difference (MCID) in subjects with shoulder pain is 2.2 cm.
Pain catastrophizing | From baseline to the end of intervention (8 weeks)
  Pain catastrophic was assessed using the Patient Catastrophizing Scale (PCS), a 52-point self-administered instrument with MCID of 4.5 points.
Kinesiophobia | From baseline to the end of intervention (8 weeks)
  Kinesiophobia was assessed using the Tampa Scale of Kinesiophobia (TSK-11), a 44-point self-administered instrument with MCID established at 6.0 points
Disability | From baseline to the end end of intervention (8 weeks)
  The degree of disability was assessed with the QuickDASH questionnaire, a self-administered instrument which expresses the degree of disability as a percentage on a scale of 0-100%, with MCID of 8% in subjects with shoulder pain.
Health-related quality of life: 5-dimension EuroQol questionnaire | From baseline to the end of intervention (8 weeks)
  The health-related quality of life was assessed with the 5-dimension EuroQol questionnaire, with MCID established on a scale of 0.03-0.52 in the population with musculoskeletal pain.

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Ponce, BSc, Principal Investigator — Universidad Santo Tomas, Chile
Locations (1):
- Hospital de Temuco, Temuco, Región de la Araucanía, Chile